CLINICAL TRIAL: NCT02624557
Title: A Phase 1, Open-label, Single-dose, Multicenter, Parallel Group Study to Assess the Pharmacokinetics and Safety of Alpelisib (BYL719) in Subjects With Hepatic Impairment Compared to Matched Healthy Control Subjects.
Brief Title: Pharmacokinetic Study of Alpelisib in Subjects With Hepatic Impairment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CBYL719A2105
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2018-05

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Healthy volunteers; Clinical pharmacology study; BYL719; alpelisib
MeSH Terms: interventions — Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate hepatic impairment group (Experimental): Subjects with moderate hepatic impairment with Child-Pugh score 7 - 9
  Interventions: Drug: Alpelisib
- Severe hepatic impairment group (Experimental): Subjects with severe hepatic impairment with Child-Pugh score 10 - 15
  Interventions: Drug: Alpelisib
- Matching healthy control group (Experimental): Subjects with apparent normal liver function matched to the hepatic impairment subjects by sex, race, age, and weight.
  Interventions: Drug: Alpelisib

INTERVENTIONS:
Drug: Alpelisib — Subjects will receive a single dose of 300 mg alpelisib.

SUMMARY:
To characterize the pharmacokinetics and safety of alpelisib in subjects with hepatic impairment compared to matched healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

-Other then hepatic impairment, subjects should be in good health as determined by past medical history, physical examination, vital signs, electrocardiogram (except for additional inclusion criteria for hepatic impaired subjects). -Subjects must weigh at least 50 kg and no more than 120 kg and have a body mass index in the range 18.0-36.0 kg/m2.

Additional criteria for hepatic impaired subjects: -Subjects must have a score clinically determined and calculated as per the Child-Pugh classification and consistent with the degree of hepatic impairment in which study is currently enrolling. -Stable Child-Pugh status within 28 days prior to dosing.

Exclusion Criteria: All subjects:

* Subject has received a liver transplant at any time in the past and is on immunosuppressant therapy.
* Smokers not willing to limit the use of tobacco to 10 cigarettes per day. -Surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject's safety in case of participation in the study. -Use of any herbal medications/supplements.

History of acute pancreatitis within 1 year of study entry.

Additional criteria for subjects with normal liver function:

-Use of any prescription or non-prescription medication. -Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.

Additional criteria for hepatic impaired subjects: -Use of any prescription or non-prescription medication, that has the potential to interact with alpelisb. Concomitant medications without potential to interact with alpelisib must be stable in dose. -Encephalopathy grade 3 or worse. -Total bilirubin > 6 mg/dl. Screening or baseline ECG: QTcF>480msec for both genders

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameter Cmax | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Measurement of effect of hepatic impairment on PK of alpelisib by assessment of the maximum plasma concentration (PK parameter Cmax). Cmax directly determined from the plasma concentration-time profile.
PK parameter AUClast | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Measurement of effect of hepatic impairment on PK of alpelisib by assessment of the PK parameter AUClast (area under the concentration-time curve from time zero to the last measurable concentration sampling time). AUC determined from the plasma concentration-time profile using non-compartmental analysis.
PK parameter AUCinf | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Measurement of effect of hepatic impairment on PK of alpelisib by assessment of the PK parameter AUCinf (area under the concentration-time curve from time zero to infinity ). AUC determined from the plasma concentration-time profile using non-compartmental analysis.

SECONDARY OUTCOMES:
PK parameter AUC0-t | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Measurement of effect of hepatic impairment on PK of alpelisib by assessment of the PK parameter AUC0-t (the partial area under the concentration-time curve from time zero to t hours post dose). AUC determined from the plasma concentration-time profile using non-compartmental analysis.
PK parameter tmax | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Measurement of effect of hepatic impairment on PK of alpelisib by assessment of the PK parameter tmax (time to reach maximum plasma concentration), directly determined from the plasma concentration-time profile.
PK parameter Cl/F | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Measurement of effect of hepatic impairment on PK of alpelisib by assessment of the PK parameter Cl/F (apparent oral total drug total plasma clearance calculated from steady-state exposure data ). Cl/F determined from the plasma concentration-time profile using non-compartmental analysis.
PK parameter Vz/F | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Measurement of effect of hepatic impairment on PK of alpelisib by assessment of the PK parameter Vz/F (the apparent volume of distribution during terminal phase). Vz/F determined from the plasma concentration-time profile using non-compartmental analysis.
PK parameter T1/2 | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Measurement of effect of hepatic impairment on PK of alpelisib by assessment of the PK parameter T1/2 (elimination half-life associated with the terminal slope (lambda-z) of a semi logarithmic concentration-time curve). T1/2 determined from the plasma concentration-time profile using non-compartmental analysis.
Relationship between PK parameters Cmax, AUClast, AUCinf and hepatic function parameters | predose, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Determination of the relationship between the primary PK parameters Cmax, AUClast, AUCinf and baseline hepatic function parameters total bilirubin, INR and serum albumin.
Adverse events severity and frequency | Baseline Day 1 to 30 days post-dose
  Assessment of safety and tolerability of a single dose alpelisib in hepatic impaired subjects compared with healthy matching control subjects by assessing the frequency and severity of adverse events based on the CTCAE criteria.
Change from baseline in laboratory parameters | Baseline Day 1 to 30 days post-dose
  Assessment of safety and tolerability of a single dose alpelisib in hepatic impaired subjects compared with healthy matching control subjects by assessing the change from baseline in hematological and biochemical laboratory parameters.
Change from baseline in ECG parameters | Baseline Day 1 to 30 days post-dose
  Assessment of safety and tolerability of a single dose alpelisib in hepatic impaired subjects compared with healthy matching control subjects by assessing the change from baseline in ECG parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - DaVita Clinical Research-Denver, Lakewood, Colorado
  - University of Miami / Clinical Research Services, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CBYL719A2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17198